CLINICAL TRIAL: NCT04698161
Title: Costituzione Della Biobanca Del Microbiota Intestinale e Salivare Umano: Dalla Disbiosi Alla Simbiosi
Brief Title: Establishment of the Human Intestinal and Salivary Microbiota Biobank - Oncologic Diseases
Acronym: BIOMIS-Onco
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Institute of Biomembranes, Bioenergetics and Molecular Biotechnologies (Other); Istituti Tumori Giovanni Paolo II (Network); University of Bari Aldo Moro (Other); University of Salento (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMIS-Onco
Record Dates: First submitted 2020-12-17; First posted 2021-01-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-01

CONDITIONS: Non Small Cell Lung Cancer; Metastatic Melanoma
Keywords: Microbioma biobank; Biological human samples; Oncologic diseases; Meta-omics approaches; Microbiota-pathology relationship
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — Surveys and Questionnaires; Independent Medical Evaluation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — faeces, saliva, blood, serum, urine, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC: Patients with non-small-cell lung cancer (NSCLC)
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- metastatic melanoma: patients with metastatic melanoma
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination

INTERVENTIONS:
Other: Biological sample collection — Collection of faeces, coproculture examination, urine, saliva, PBMC and blood for biobanking, to evaluate the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile, and to perform routine screening. Analysis for the identification, quantification and characterization of health-promoting bacteria
Other: Questionnaire — Anamnestic questionnaire, 3-day food questionnaire, Food Frequency Questionnaire
Other: Medical examination — Blood pressure measurement, abdominal and thoracic physical examination

SUMMARY:
This is a prospective, clinical, multicentre study aimed to collect biological samples and study microbiota from subjects with non-small-cell lung cancer (NSCLC) and metastatic melanoma. Microbiota is a complex consortium of microorganisms, located at the mucosal level (in particular intestinal, oral and vaginal) having a key role in human health and in the onset of several diseases. Microbiota alterations have been found in several diseases (gastrointestinal, metabolic, renal, oncological, gynaecological)

The study will allow to:

* Provide biological samples (faeces, saliva, blood, urine) from oncologic patients to the first Italian microbiota biobank;
* Study microorganisms using different in vitro and in vivo techniques;
* Study the link between the microbiota and the disease. This study is part of the BIOMIS project (Project Code: ARS01_01220), presented as part of the "Avviso per la presentazione di progetti di ricerca industriale e sviluppo sperimentale nelle 12 aree di specializzazione individuate dal PNR 2015-2020" and admitted to funding under the National Operational Program "Ricerca e Innovazione" 2014-2020 by directorial decree of MIUR - Department for Higher Education and Research - n. 2298 of 12 September 2018. BIOMIS includes several clinical studies that enrol patients with different pathologies to collect and store biological samples and study microbiota.

DETAILED DESCRIPTION:
The primary aim of this multicentric study is to populate the first national microbioma biobank with biological samples (fecal, salivary, urinary and blood samples) subjects suffering from selected oncologic diseases, i.e. non-small-cell lung cancer (NSCLC) and metastatic melanoma. The secondary aim is the characterization of microorganisms of the biobank and study of the microbiota-pathology relationship using meta-omics, in vitro and in vivo approaches.

The study plans to enrol 50 subjects at IRCCSS Istituto Tumori di Bari, according to the inclusion/exclusion criteria. The study participation is voluntary, and the subjects have the right to withdraw from the study at any time and for any reason.

During the study, 3 visits are planned:

* Visit 0 (V0), including description of the objectives and procedures study, signature written informed consent, inclusion/exclusion criteria evaluation, medical examination (blood pressure measurement, abdominal and thoracic physical examination), filling in of the anamnestic questionnaire, delivery of the coproculture kit, delivery of kits for the collection of fecal, salivary and urinary material to be reported at Visit 1 and delivery of a 3-day food diary, to be completed autonomously in the days preceding the Visit 1.
* Visit 1 (V1) - delivery of the of the collected biological material (feces, saliva, urine), and of a 3-day food diary, filling in of the new signs and symptoms anamnestic questionnaire and blood sampling by medical staff.
* Telephone evaluation: administration of a "Food Frequency Questionnaire" to assess the subjects' alimentary habits.

Standard Operative Procedures (SOP) for samples storing, transport and processing will be adopted to ensure samples stability and grant results validity and quality.

Following collections, samples will be processed in different aliquots that will be used for:

* routine screening;
* storage in the I.R.C.C.S. - Istituto Tumori "Giovanni Paolo II" human microbiote biobank;
* evaluation of the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile;
* Evaluation of the transcriptomic profile of PBMCs of healthy subjects and subjects affected by selected pathologies and evaluation of the serum proteomic profile Furthermore, molecular characterization of pathogenic microorganisms and pathogenic biotypes (pathovars) of commensal species of subjects with selected pathologies will be conducted.

Part of the biological material will be used for animal studies on the physiopathological role of the human intestinal microbiota transplanted into mouse models of pathology and Germ-free mouse models (specific animal study protocol developed).

Also, in vitro studies on mucosal models to evaluate the interaction between the microbiota and the intestinal mucosa will be conducted.

The study foresees no more than minimal risk associated with blood sampling procedures. All the necessary measures to avoid any risks / inconveniences resulting from participation of the subject under study will be taken.

The study is compliant with Good Clinical Practice. Study protocol and all related documents have been approved by approved by the Independent Ethics Committees (IEC) of the involved clinical sites.

To ensure the protection and confidentiality of the participants' data, all study activities will be carried out in accordance with the European General Data Protection Regulation, Regulation (EU) 2016/679, which repeals Directive 95/46/EC.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS WITH NSLSC

* NSLSC diagnosis
* aged between 18 and 75 years
* omnivorous diet
* having suspended antibiotic therapy for at least 15 days
* cessation of treatment with cortisone for at least 15 days
* signature of the informed consent

PATIENTS WITH METASTATIC MELANOMA

* metastatic melanoma diagnosis
* aged between 18 and 75 years
* omnivorous diet
* having suspended antibiotic therapy for at least 15 days
* cessation of treatment with cortisone for at least 15 days
* signature of the informed consent

Exclusion Criteria:

PATIENTS WITH NSLSC/METASTATIC MELANOMA

Exclusion criteria:

* Current treatment with antibiotics or immunosuppressive drugs Previous chemotherapy treatmment Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent onset of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* Hypertension
* eGFR (estimated glomerular filtration rate) lower than 60ml / minute and / or diagnosis of nephropathy
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Psychiatric conditions that reduce protocol compliance.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with non-small-cell lung cancer (NSCLC) and metastatic melanoma attending the IRCSS Istituto Tumori di Bari. Enrolled subjects must not have any family relationship and hierarchical subordination with the hospitals in which biological samples will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Biological samples collection for establishment of the first National Microbiome Biobank | through study completion, an average of 1 year
  Recruitment of 50 subjects (non-small-cell lung cancer and metastatic melanoma patients) to collect biological samples for establishment of the first National Microbiome Biobank

CONTACTS AND LOCATIONS:
Overall Officials: Angelo V Paradiso, MD, Principal Investigator — IRCCS Istituto Tumori Giovanni Paolo II
Locations (1):
- IRCCS Istituto Tumori Giovanni Paolo II, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bingula R, Filaire M, Radosevic-Robin N, Berthon JY, Bernalier-Donadille A, Vasson MP, Thivat E, Kwiatkowski F, Filaire E. Characterisation of gut, lung, and upper airways microbiota in patients with non-small cell lung carcinoma: Study protocol for case-control observational trial. Medicine (Baltimore). 2018 Dec;97(50):e13676. doi: 10.1097/MD.0000000000013676. PMID 30558074
- [Background] Matson V, Fessler J, Bao R, Chongsuwat T, Zha Y, Alegre ML, Luke JJ, Gajewski TF. The commensal microbiome is associated with anti-PD-1 efficacy in metastatic melanoma patients. Science. 2018 Jan 5;359(6371):104-108. doi: 10.1126/science.aao3290. PMID 29302014
- [Background] Frankel AE, Coughlin LA, Kim J, Froehlich TW, Xie Y, Frenkel EP, Koh AY. Metagenomic Shotgun Sequencing and Unbiased Metabolomic Profiling Identify Specific Human Gut Microbiota and Metabolites Associated with Immune Checkpoint Therapy Efficacy in Melanoma Patients. Neoplasia. 2017 Oct;19(10):848-855. doi: 10.1016/j.neo.2017.08.004. Epub 2017 Sep 15. PMID 28923537
- [Background] Chaput N, Lepage P, Coutzac C, Soularue E, Le Roux K, Monot C, Boselli L, Routier E, Cassard L, Collins M, Vaysse T, Marthey L, Eggermont A, Asvatourian V, Lanoy E, Mateus C, Robert C, Carbonnel F. Baseline gut microbiota predicts clinical response and colitis in metastatic melanoma patients treated with ipilimumab. Ann Oncol. 2017 Jun 1;28(6):1368-1379. doi: 10.1093/annonc/mdx108. PMID 28368458
- [Background] Dubin K, Callahan MK, Ren B, Khanin R, Viale A, Ling L, No D, Gobourne A, Littmann E, Huttenhower C, Pamer EG, Wolchok JD. Intestinal microbiome analyses identify melanoma patients at risk for checkpoint-blockade-induced colitis. Nat Commun. 2016 Feb 2;7:10391. doi: 10.1038/ncomms10391. PMID 26837003